CLINICAL TRIAL: NCT01474655
Title: Assessment of Retinal Layers and Visual Rehabilitation After Epiretinal Membrane Removal
Brief Title: Retinal Layers and Visual Rehabilitation After Epiretinal Membrane Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Se Woong, Kang, Professor, Samsung Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011-07-069
Record Dates: First submitted 2011-10-21; First posted 2011-11-18 (Estimated); Last update posted 2011-11-18 (Estimated); Status verified 2011-11

CONDITIONS: Epiretinal Membrane
Keywords: epiretinal membrane; visual acuity; metamorphopsia; thickness of retinal layers; spectral domain optical coherence tomography
MeSH Terms: conditions — Epiretinal Membrane; Vision Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Pars plana vitrectomy and removal of epiretinal membrane — A three-port standard pars plana vitrectomy was performed by a single surgeon using a 23-gauge vitrectomy system, either Associate®(Dutch Ophthalmic Research Center. Inc., Zuidland, The Netherlands) or Accurus®(Alcon Laboratories Inc., Fort Worth, USA), with one step scleral tunnel incision. Visualization of the fundus was achieved using a wide-angle viewing system. After core vitrectomy, induction of a posterior vitreous detachment was conducted using a 23-gauge angulated dissecting needle in cases without presence of a posterior vitreous detachment. The epiretinal membrane and internal limiting membrane was removed in all eyes. In most cases, internal limiting membrane was removed without the assistance of staining dye. Indocyanine green dye was used to facilitate the removal of internal limiting membrane in some of the cases.

SUMMARY:
The purpose of this study is to evaluate the changes in visual acuity, metamorphopsia, and thickness of retinal layers after epiretinal membrane removal and to investigate factors associated with visual function.

DETAILED DESCRIPTION:
Eyes with idiopathic Epiretinal Membrane Removal (ERM) scheduled to underwent ERM removal were included. Changes in visual acuity, metamorphopsia score (M-score) using M-chart, and parafoveal thickness of each retinal layer were evaluated preoperatively and at 2-month and 6-month postoperative follow-up visits. Factors associated with visual acuity and M-score were investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed with idiopathic epiretinal membrane and were scheduled for epiretinal membrane removal

Exclusion Criteria:

* evidence of ocular inflammation, diabetic retinopathy, hypertensive retinopathy, and retinal vasculitis, media opacity that would influence visual acuity or preclude acquisition of clear spectral domain optical coherence tomography images,
* presence of cataract judged to affect visual function, -6.0 diopters or more of spherical equivalent, prominent staphyloma, history of intraocular surgery other than uncomplicated cataract surgery, history of retinal detachment, other ocular diseases that may influence the macular microstructure or visual function, immeasurable fovea location on the spectral domain optical coherence tomography image due to severe retinal contraction, and indistinct intraretinal structure on spectral domain optical coherence tomography images.
* patients who underwent combined epiretinal membrane removal and cataract extraction, less than six months follow-up after epiretinal membrane removal, who had occurrence or progression of cataract after the surgery judged to affect visual function, or who experienced recurrence of epiretinal membrane during the follow-up period

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-09; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Postoperative changes in visual acuity | preop, 2-month postop, 6-months postop
  Changes in visual acuity (Early treatment diabetic retinopathy study score)was evaluated preoperatively and at 2-month and 6-month postoperative follow-up visits.
Postoperative changes in metamorphopsia | preop, 2 months postop, 6 months postop
  Changes in metamorphopsia score (M-score) was measured using M-chart and evaluated preoperatively and at 2-month and 6-month postoperative follow-up visits.
Postoperative parafoveal thickness of each retinal layer | preop, 2 months postop, 6 months postop
  Changes in parafoveal thickness of each retinal layer was evaluated based on spectral domain optical coherence tomography images

CONTACTS AND LOCATIONS:
Overall Officials: Se Woong Kang, M.D., Principal Investigator — Department of Ophthalmology, Samsung Medical Center, Sungkyunkwan University School of Medicine

REFERENCES:
- [Derived] Kim JH, Kang SW, Kong MG, Ha HS. Assessment of retinal layers and visual rehabilitation after epiretinal membrane removal. Graefes Arch Clin Exp Ophthalmol. 2013 Apr;251(4):1055-64. doi: 10.1007/s00417-012-2120-7. Epub 2012 Aug 9. PMID 22875136